CLINICAL TRIAL: NCT05532800
Title: A Randomized, Double-blind, Placebo-controlled Phase III Clinical Study Evaluating the Efficacy and Safety of JS002 Prefilled Syringes(PFS) and Prefilled Autosyringes(AI) in Patients With Primary Hypercholesterolemia and Mixed Hyperlipidemia
Brief Title: The Efficacy and Safety of JS002 PFS and AI in Patients With Primary Hypercholesterolemia and Mixed Hyperlipidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JS002-006
Record Dates: First submitted 2022-09-05; First posted 2022-09-08 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Hyperlipemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JS002 (Experimental): Cobort 1:150 mg/1mL Q2W PFS,Cobort 2:150 mg/1mL Q2W AI
  Interventions: Drug: JS002
- Placebo (Placebo Comparator): Cobort 1:/1mL Q2W PFS,Cobort 2:1mL Q2W AI
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JS002 — JS002:150mg(1mL) Q2W PFS, Placebo: 1mL Q2W PFS.
  Arms: JS002
Drug: Placebo — JS002:150mg(1mL) Q2W AI, Placebo: 1mL Q2W AI.
  Arms: Placebo

SUMMARY:
JS002 is a recombinant humanized anti-PCSK9 monoclonal antibody. This is a randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of JS002 prefilled syringes and prefilled autosyringes in patients with primary hypercholesterolemia and mixed hyperlipidemia when combined with statin therapy.

In this study, one dose group (150 mg) were set up in this study. 240 subjects are plan to be enrolled (the study drug will be assigned to a 2:1 :2:1ratio of JS002 PFS / placebo or JS002 AI / placebo ).

Each subject required a maximum of 6 weeks of screening, 12 weeks of treatment, and 8 weeks of follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Age 18~80 years old;
3. Stable optimized LLT at least 4 weeks before randomization;
4. Two times of Fasting triglycerides ≤4.5 mmol/L(400mg/dL)at the time of screening;

Exclusion Criteria:

1. History of NYHA class III-IV heart failure or EF<30%;
2. History of uncontrolled arrhythmia within 90 days;
3. History of MI,UA, PCI or CABG, stroke within 90 days;
4. Known hemorrhagic stroke disease;
5. Planned cardiac surgery or revascularization.
6. Uncontrolled hypertension.
7. Uncontrolled diabetes mellitius (HbA1c>8.0%）.
8. Other conditions that the researchers considered inappropriate to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2023-02-09 (Actual)

PRIMARY OUTCOMES:
LDL-C with JS002 PFS | at week 12
  Percentage change in LDL-C relative to baseline at Week 12 with JS002 PFS
LDL-C with JS002 AI | at week 12
  Percentage change in LDL-C relative to baseline at Week 12 with JS002 AI

SECONDARY OUTCOMES:
LDL-C with JS002 PFS | at week 12
  The absolute change in LDL-C relative to baseline with JS002 PFS
LDL-C with JS002 AI | at week 12
  The absolute change in LDL-C relative to baseline with JS002 AI
lipid parameters | at week 12
  Percentages and absolute change in other lipid parameters to baseline with JS002 PFS and JS002 AI
LDL-C reduction≥50 with JS002 PFS | at week 12
  Proportion of subjects with a ≥50% reduction in serum LDL-C at 12 weeks after subcutaneous treatment with JS002 PFS from baseline
LDL-C reduction≥50 with JS002 AI | at week 12
  Proportion of subjects with a ≥50% reduction in serum LDL-C at 12 weeks after subcutaneous treatment with JS002 AI from baseline
LDL-C dropped to < 70 mg/dL with JS002 PFS | at week 12
  Proportion of subjects whose serum LDL-C dropped to < 70 mg/dL (1.8 mmol/L) at 12 weeks after subcutaneous injection of JS002 PFS
LDL-C dropped to < 70 mg/dL with JS002 AI | at week 12
  Proportion of subjects whose serum LDL-C dropped to < 70 mg/dL (1.8 mmol/L) at 12 weeks after subcutaneous injection of JS002 AI
full dose | at week 0, 2, 4, 6, 8, 10
  Proportion of subjects receiving full dose of JS002 AI during treatment (weeks 0, 2, 4, 6, 8, 10)

CONTACTS AND LOCATIONS:
Locations (21):
- China (21):
  - Beijing Anzhen Hospital，Capital Medical University, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Daqing People's Hospital, Daqing, Heilongjiang
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Jingzhou Central Hospital, Jingzhou, Hubei
  - The Second Xiangya Hospital Of Central South University, Changsha, Hunan
  - Changzhou Second People's Hospital, Changzhou, Jiangsu
  - Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Nanchang First Hospital, Nanchang, Jiangxi
  - Nanchang Third Hospital, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Dalian Municipal Central Hospital, Dalian, Liaoning
  - The First Affiliated Hospital of Jinzhou Medical University, Jinzhou, Liaoning
  - Xianyang Hospital of Yan'an University, Xianyang, Shanxi
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality
  - Taizhou Hospital Of Zhejiang Province, Taizhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No